CLINICAL TRIAL: NCT02361294
Title: Prospective Study to Generate Hypotheses About the Role of Platelets and Immature Platelets in the Pathogenesis of Idiopathic Venous Thromboses and Pulmonary Embolisms
Brief Title: Immature Plateletes in the Etiopathology of Deep Venous Thrombosis
Acronym: iPLATELET
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: TechnischeUM 1
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Immature Platelets; Deep Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — thrombophilia screening
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient: Patients with a newly diagnosed deep venous thrombosis and/or pulmonary embolism. The thrombembolism is idiopathic or caused by immobilisation. Three blood samples are taken during the study period. A thrombophilia screening is carried out.
  Interventions: Other: Blood samples
- Control: Patients that present with a suspicion of deep venous thrombosis which is excluded by duplex sonography. One to two blood samples are taken during the study period.
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples

SUMMARY:
The study is designed to evaluate the role of platelets and immature platelets in the ethiopathology of deep venous thrombosis and pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a newly diagnosed deep venous thrombosis and/or pulmonary embolism. The thrombembolism is idiopathic or caused by immobilisation.
* Control: Patients that present with a suspicion of deep venous thrombosis which is excluded by duplex sonography.

Exclusion Criteria:

* therapy with glycoprotein IIb/IIIa-antagonists within the last 10 days
* therapy with antiplatelet drugs (ASA, Clopidogrel, Ticagrelor, Prasugrel, Dipyridamol)
* preexisting anticoagulation
* number of platelets < 100.000/µl
* anemia (hematocrit < 35%, Hb < 10 g/dl)
* age > 80 y or < 18 y
* renal insufficiency GFR < 30 ml/min
* hepatic impairment with an increased risk for bleeding or coagulopathy, or liver cirrhosis (≥ Child Pugh B)
* intracranial or intracerebral bleeding within the last six months
* intraspinal or intracerebral vascular anomalies
* clinically relevant acute bleedings
* malign disease
* infections within the last 7 d
* hematological, rheumatologic and autoimmune diseases
* operations within the last six months
* transfusion of rec celll concentrates within the last six months
* transfusion of fresh frozen plasma or platelet concentrates within the last month
* preexisting medication with CYP 3A4 inhibitors and inductors, p-glycoprotein inhibitors (Azol-Antimycotis, HIV protease-inhibitors)
* hypersensitivity/contraindications for Rivaroxaban
* pregnancy or lactation
* thrombophilia
* thrombocytopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all-comers
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2014-12; Primary Completion 2017-04-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Significantly increased proportion of immature platelets in patients with deep venous thrombosis and/or pulmonary embolism compared to the control. | at time of diagnosis

SECONDARY OUTCOMES:
Significantly higher values of platelet function in patients with deep venous thrombosis and/or pulmonary embolism compared to the control. | at time of diagnosis
A persistently increased proportion of immature platelets in patients with deep venous thrombosis and/or pulmonary embolism compared to the controls three months after diagnosis. | 3 months after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Tareq Ibrahim, MD, Principal Investigator — Senior consultant
Locations (1):
- Klinikum rechts der Isar, Technische Universität München, Munich, Germany